CLINICAL TRIAL: NCT00824356
Title: A Randomised, Double-Blind, Placebo-Controlled, 3-Period Crossover Study to Assess the Efficacy and Safety of Single Dose Intranasal GSK1004723 Compared With Placebo in an Allergen Challenge Chamber in Male Subjects With Seasonal Allergic Rhinitis
Brief Title: Allergen Challenge Chamber Study With Single Dose Intranasal GSK1004723 Compared With Placebo
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 110159; 723 PoC
Record Dates: First submitted 2009-01-08; First posted 2009-01-16 (Estimated); Last update posted 2009-06-22 (Estimated); Status verified 2009-06

CONDITIONS: Allergic Rhinitis
Keywords: Allergic Rhinitis; Proof-of-Concept
MeSH Terms: conditions — Rhinitis, Allergic | interventions — GSK 1004723

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (3):
- GSK1004726 (1000mg) (Active Comparator): 1000mg aqueous suspension
  Interventions: Drug: GSK1004723 (1000mg)
- Placebo (Placebo Comparator): Intranasal spray
  Interventions: Other: Placebo; Drug: GSK1004723 (1000mg)
- GSK1004723 (200mg) (Active Comparator): 200 mg aqueous suspension
  Interventions: Drug: GSK1004723 (200mg)

INTERVENTIONS:
Drug: GSK1004723 (200mg) — Intranasal antihistamine.
  Arms: GSK1004723 (200mg)
Other: Placebo — Equivalent to GSK1004723 in presentation etc.
  Arms: Placebo
Drug: GSK1004723 (1000mg) — Intranasal antihistamine.
  Arms: GSK1004726 (1000mg); Placebo

SUMMARY:
This is a placebo-controlled, 3-period crossover study to assess the efficacy and safety of two single doses of an intranasal anti-histamine GSK1004723 compared with placebo in an allergen challenge chamber in male subjects with seasonal allergic

ELIGIBILITY:
Inclusion Criteria:

* Subject is healthy apart from seasonal allergic rhinitis, as determined by a physician. Can have mild asthma.
* Male
* Aged 18 - 65
* Weight 50kg+, BMI 19-32 kg/m2
* Exhibit response to Challenge Chamber and skin prick test.
* Non-smoker
* Capable of giving informed consent

Exclusion Criteria:

* No nasal structural abnornmality/polyposis, surgery, infection.
* any respiratory disease, other than mild asthma or seasonal allergic rhinitis
* participated in another clinical study within 30 days.
* Subject has donated a unit of blood within 1 month
* Use of prescription or non-prescription drugs, including vitamins and st john's wort within 7 days of trial.
* History of sensitivty to drug
* History of alcohol/drug abuse within 12 months.
* Positive Hepatitis B antibody test
* Positive HIV antibody test
* Risk of non-compliance with study protocol
* Perenial allergic rhinitis
* Administration of oral, injectable or dermal corticosteriods within 8 weeks, intranasal or inhaled within 3 weeks.
* Past or present disease that may affect outcome, as judge by investigator Specific Immunotherapy within 2 years

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2008-06; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in total nasal symptom score 0-4 hours post dose | 0-4 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Hanover, Lower Saxony, Germany